CLINICAL TRIAL: NCT05979493
Title: Quadratus Lumborum Block to Improve Postoperative Pain Management After Laparoscopic Myomectomies: a Double-blinded and Prospective Randomized Clinical Trial.
Brief Title: QL Block in Laparoscopic Myomectomy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Joseph Findley MD (Other)
Responsible Party: Sponsor-Investigator, Joseph Findley MD, University Hospitals Department of Reproductive Endocrinology and Infertility, University Hospitals Cleveland Medical Center
Organization: University Hospitals Cleveland Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: STUDY20230830
Record Dates: First submitted 2023-07-28; First posted 2023-08-07 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Postoperative Pain; Fibroid Uterus
Keywords: QL Block; Myomectomy
MeSH Terms: conditions — Pain, Postoperative; Leiomyoma | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- QL Block with Bupivacaine (Experimental): Participants will get a QL block using 30cc Bupivacaine bilaterally in quadratus lumborum muscle (60cc total).
  Interventions: Drug: Bupivacain
- Control (Sham Comparator): Participants will get a sham injection of 30cc saline bilaterally in quadratus lumborum muscle (60cc total).
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Bupivacain — 30cc IM injection in each quadratus lumborum muscle (60cc total).
  Arms: QL Block with Bupivacaine
Drug: Saline — 30cc IM injection in each quadratus lumborum muscle (60cc total).
  Arms: Control

SUMMARY:
This study aims to determine the efficacy of a quadratus lumborum (QL) block in decreasing postoperative pain in patients undergoing myomectomy for uterine fibroids. A QL block is a temporary anesthetic injection in the quadratus lumborum muscle, a muscle in the lower back, that has been previously shown to significantly reduce postoperative pain levels in patients undergoing abdominal and pelvic surgery. Because of its demonstrated effects, the QL block is becoming a standard of anesthesia and surgical care. Since participants will be undergoing a myomectomy procedure, the investigators believe that participants may qualify to participate in this study. The investigators will be comparing patients who receive the QL block (in addition to standard anesthesia and postoperative pain care) with patients who do not receive the QL block (in addition to standard care). The participants will be randomly assigned to one of the two groups and may or may not actually receive the block.

ELIGIBILITY:
Inclusion Criteria:

* Presence of uterine fibroids requiring surgical excision with preservation of the uterus
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Provision of signed and dated informed consent form

Exclusion Criteria:

* Pre-existing diagnoses of anxiety or depression
* Pre-existing coagulopathies
* Pre-existing neuropathic or chronic pelvic pain
* Chronic opioid use
* Illiteracy due to inability to read and understand plain questionnaire
* Non-English speaking
* BMI >38

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2024-08-24 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-03 (Estimated)

PRIMARY OUTCOMES:
Time in minutes from first analgesic request as measured by medical chart review | Up to 24 hours
Total number of doses of rescue analgesics given as measured by medical chart review | Up to 24 hours

SECONDARY OUTCOMES:
Pain as measured by visual analog scale (VAS) | Up to 48 hours after discharge from hospital.
  VAS is a pain scale from 0-10 with 0 being no pain and 10 being the worst pain ever.
Patient satisfaction with perioperative pain management measured on a scale of 1-10 | Up to 48 hours after discharge from hospital.
  Pain management scale with 1 being very disappointed in pain management with 10 being highly satisfied with pain managment.

OTHER OUTCOMES:
Pain as measured by Richmond Agitation Sedation Scale (RASS) | Up to 24 hours
  RASS is measured from -5 to +4 with -5 being no response to voice or physical stimulation and +4 being overtly combative, violent, immediate danger to staff

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Findley, MD, Principal Investigator — University Hospitals
Locations (1):
- University Hospitals Ahuja Medical Center, Beachwood, Ohio, United States

IPD SHARING:
Plan to Share IPD: No